CLINICAL TRIAL: NCT02018627
Title: Equivalence of A Stable Liquid Glucagon Formulation With Freshly Reconstituted Lyophilized Glucagon
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Steven J. Russell, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002549
Record Dates: First submitted 2013-12-16; First posted 2013-12-23 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Type 1 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xeris glucagon (Experimental): Xeris glucagon 50 micrograms, subcutaneous injection
  Interventions: Drug: Xeris glucagon
- Lilly glucagon (Active Comparator): Lilly glucagon 30 micrograms, subcutaneous injection
  Interventions: Drug: Lilly glucagon

INTERVENTIONS:
Drug: Xeris glucagon — The subject is given an injection of xeris glucagon
  Arms: Xeris glucagon
Drug: Lilly glucagon — The subject is given an injection of lilly glucagon
  Arms: Lilly glucagon

SUMMARY:
This study will test the hypothesis that micro-doses of Xerisol Glucagon (Xeris Pharmaceuticals) will be non-inferior by pharmacokinetic and pharmacodynamic criteria vs. micro-doses of Glucagon for Injection (Eli Lilly).

DETAILED DESCRIPTION:
This study will test the hypothesis that micro-doses of a new formulation of stable glucagon, Xerisol Glucagon (Xeris Pharmaceuticals), will be non-inferior by pharmacokinetic and pharmacodynamic criteria vs. micro-doses of a freshly reconstituted formulation of glucagon that has poor stability in solution, Glucagon for Injection (Eli Lilly).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 80 years old with type 1 diabetes for at least one year.
* Diabetes managed using an insulin infusion pump using rapid-acting insulin such as insulin aspart (NovoLog), insulin lispro (Humalog), and insulin glulisine (Apidra) for at least one week prior to enrollment.

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to comply with study procedures.
* Current participation in another diabetes-related clinical trial that, in the judgment of the principle investigator, will compromise the results of the clamp study or the safety of the subject.
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception.
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
* Hemoglobin < 11.5 gm/dl.
* History of pheochromocytoma. Fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor (paroxysms of tachycardia, pallor, or headache; personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease; episodic or treatment of refractory hypertension, defined as requiring 4 or more medications to achieve normotension).
* History of adverse reaction to glucagon (including allergy) besides nausea, vomiting, or headache.
* Inadequate venous access as determined by study nurse or physician at time of screening.
* Liver failure or cirrhosis.
* Any other factors that, in the judgment of the principal investigator, would interfere with the safe completion of the study procedures.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 subjects were enrolled in this study. One was ineligible after enrollment. 4 were enrolled and eligible, but were not able to schedule their study visit. 2 participated in "test run" experiments as we adjusted glucagon doses to account for concentration differences. 13 subjects completed experiments using the same protocol.
Groups:
- Xeris Glucagon First, Then Lilly Glucagon: Xeris glucagon 50 micrograms, subcutaneous injection then Lilly glucagon 30 micrograms, subcutaneous injection
  Lilly glucagon: The subject is given an injection of lilly glucagon Xeris glucagon: The subject is given an injection of xeris glucagon
- Lilly Glucagon First, Then Xeris Glucagon: Lilly glucagon 30 micrograms, subcutaneous injection then Xeris glucagon 50 micrograms, subcutaneous injection
  Lilly glucagon: The subject is given an injection of lilly glucagon Xeris glucagon: The subject is given an injection of xeris glucagon
Period: Overall Study
Arm/Group | Xeris Glucagon First, Then Lilly Glucagon | Lilly Glucagon First, Then Xeris Glucagon
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Xeris Glucagon First, Then Lilly Glucagon: Xeris glucagon 50 micrograms, subcutaneous injection, then Lilly glucagon 30 micrograms, subcutaneous injection
  Xeris glucagon: The subject is given an injection of xeris glucagon Lilly glucagon: The subject is given an injection of lilly glucagon
- Lilly Glucagon First, Then Xeris Glucagon: Lilly glucagon 30 micrograms, subcutaneous injection, then Xeris glucagon 50 micrograms, subcutaneous injection
  Lilly glucagon: The subject is given an injection of lilly glucagon Xeris glucagon: The subject is given an injection of xeris glucagon
- Total: Total of all reporting groups
Arm/Group | Xeris Glucagon First, Then Lilly Glucagon | Lilly Glucagon First, Then Xeris Glucagon | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (11.8) | 45.6 (11.9) | 51.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 1 | 0 | 1
Hemoglobin A1c [Mean (Standard Deviation); unit: percent] | 7.4 (1.3) | 7.0 (0.6) | 7.2 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Tmax
Description: tmax for Xeris vs. Lilly (non-inferiority)
Time Frame: every 2 minutes for 1 hour post-dose of each glucagon
Population: 13 subjects completed the study following a consistent protocol using the glucagon doses described in the arm/group description. 7 subjects were randomized to get Xeris glucagon first, 6 subjects were randomized to get Lilly glucagon first. All 13 subjects received both glucagon injections, and the data is reported for each drug.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
minutes | 23.8 (9.3) | 15.7 (3.0)

2. Secondary Outcome: AOCGIR
Description: Area over the curve for glucose infusion rate in the hour following administration (AOCGIR) for Xeris vs. Lilly (non-inferiority)
Time Frame: every 2 minutes for 1 hour post-dose of each glucagon
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*min/kg
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
mg*min/kg | 201.1 (275.5) | 132.2 (87.9)

3. Secondary Outcome: GIRmin
Description: Minimal glucose infusion rate (GIRmin) for Xeris vs. Lilly (non-inferiority)
Time Frame: every 2 minutes for 1 hour post-dose of each glucagon
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dextrose mg/kg/min
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
dextrose mg/kg/min | 2.9 (2.2) | 2.9 (1.8)

4. Secondary Outcome: t½Max
Description: Glucagon t½max for Xeris vs. Lilly (non-inferiority)
Time Frame: every 2 minutes for 1 hour post-dose of each glucagon
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
minutes | 11.3 (3.1) | 5.9 (2.1)

5. Secondary Outcome: Injection Pain
Description: Quantitation of adverse events related to glucagon injection for Xeris vs. Lilly:
  -average Injection pain on a 10 cm standard VAS: 0 = no pain, 10 = worst imaginable pain reported immediately after injection of glucagon
Time Frame: immediately after injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
cm | 13.8 (17.7) | 7.6 (8.7)

6. Secondary Outcome: Injection Site Erythema
Description: Quantitation of adverse events related to glucagon injection for Xeris vs. Lilly:
  -Injection site erythema or other local reaction, maximum diameter within 1 hour of injection
Time Frame: within 1 hour of injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
cm | 0 (0) | 0 (0)

7. Secondary Outcome: Maximal Nausea
Description: Quantitation of adverse events related to glucagon injection for Xeris vs. Lilly:
  -Maximal nausea within 1 hour of injection on a 10 cm VAS: no nausea = 0, vomiting = 10
Time Frame: within 1 hour of injection
Population: as for outcome 1
Measure: Number; unit: cm
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
cm | 1.0 | 2.3

8. Secondary Outcome: Dermal Response (Draize Scale for Erythema and Eschar Formation)
Description: Average grade on the erythema and eschar formation portion of the Draize scale for dermal response (0 being the lowest, 4 being the highest)
Time Frame: within 1 hour of injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on draize scale
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
score on draize scale | 0 (0) | 0 (0)

9. Secondary Outcome: Dermal Response (Draize Scale Grade for Edema Formation)
Description: Average grade on the edema formation portion of the Draize scale for dermal response (0 being the lowest, 4 being the highest)
Time Frame: within 1 hour of injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on draize scale
Arm/Group | Xeris Glucagon | Lilly Glucagon
Number analyzed (Participants) | 13 | 13
score on draize scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Xeris Glucagon | Lilly Glucagon
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT02018627/Prot_SAP_000.pdf